CLINICAL TRIAL: NCT03759223
Title: Enhanced Problem-Solving Training (E-PST) to Improve Recovery From mTBI
Brief Title: Enhanced Problem-Solving Training
Acronym: E-PST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2796-W; RX002796 (Other Grant/Funding Number: VA Rehabilitation Research & Development (RR&D))
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Brain Concussion
Keywords: Mild Traumatic Brain Injury; Concussion, Mild; Veterans; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Up to 12 participants will first complete an open trial of E-PST to test the feasibility, acceptability, and preliminary clinical effect. Subsequently, up to 38 participants will be randomly assigned (1:1) to E-PST or a control condition comprised of supportive contact and symptom monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- E-PST (randomized) (Experimental): Enhanced Problem-Solving Training (E-PST) arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Randomized participants were assigned 1:1 to E-PST or HLM.
  Interventions: Behavioral: Enhanced Problem-Solving Training (E-PST)
- Control (randomized) (Active Comparator): Healthy Living Messages (Control) arm. Healthy Living Messages (HLM) are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care. Randomized participants were assigned 1:1 to E-PST or HLM.
  Interventions: Behavioral: Healthy Living Messages (HLM)
- E-PST (non-randomized) (Other): Enhanced Problem-Solving Training (E-PST) arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Non-randomized participants were assigned to E-PST only.
  Interventions: Behavioral: Enhanced Problem-Solving Training (E-PST) (non-randomized)

INTERVENTIONS:
Behavioral: Enhanced Problem-Solving Training (E-PST) — E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Randomized participants were assigned 1:1 to E-PST or HLM.
  Other Names: Problem-Solving Training for Concussion (PST-Concussion)
  Arms: E-PST (randomized)
Behavioral: Healthy Living Messages (HLM) — Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care. Randomized participants were assigned 1:1 to E-PST or HLM.
  Other Names: Control
  Arms: Control (randomized)
Behavioral: Enhanced Problem-Solving Training (E-PST) (non-randomized) — E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Non-randomized participants were assigned to E-PST only.
  Other Names: Problem-Solving Training for Concussion (PST-Concussion)
  Arms: E-PST (non-randomized)

SUMMARY:
Mild traumatic brain injury (mTBI) is among the most common injuries sustained by Veterans of Operations Enduring and Iraqi Freedom. It is also highly co-morbid with mental health conditions, such as post-traumatic stress disorder and depression. While mTBI alone is not typically thought to cause lasting deficits in personal functioning or cognitive abilities, Veterans with a history of mTBI nonetheless report chronic psychological distress, as well as subjective difficulties with attention, concentration, poor frustration tolerance, and decision-making. Although current clinical practice guidelines for mTBI emphasize primary care-based symptom management, there are presently no evidence-based interventions to treat mental health symptoms in this setting. This research proposal therefore seeks to adapt and pilot test a brief, primary care-based intervention (E-PST) to reduce psychological distress in Veterans with mTBI by augmenting problem-solving skills, and helping them to develop specific cognitive and behavioral skills to improve upon their self-reported cognitive inefficiencies. The investigators hypothesize that Veterans who complete E-PST will report improvements in psychological distress compared to participants in the control condition.

DETAILED DESCRIPTION:
Open Trial: The primary focus of the open trial is to gather feasibility and acceptability data from up to 12 participants, though clinical effect will also be evaluated using select measures outlined below. Feasibility metrics will be internally monitored. Participant feedback on the acceptability of E-PST will be gathered following each treatment session. Qualitative data will be analyzed using rapid qualitative analysis. Given the small sample, clinical effect will be descriptively explored. Individual line graphs of pre-post Brief Symptom Inventory-18 (BSI-18) scores will be generated, and mean differences in BSI-18 scores will be compared. Trends in change scores will be visually inspected to evaluate evidence of a preliminary clinical effect.

Randomized Trial: The focus of the randomized trial is threefold: a) to estimate a preliminary effect size for the primary outcome measure (BSI-18); b) determine the feasibility of the assessment plan; and c) establish feasibility of recruitment and retention in order to guide the design of a future multi-site efficacy trial. BSI-18 data will be described with means, standard deviations, and confidence intervals at each time point and condition. To show central tendency, variation and potential trends over time, means and 95% confidence intervals will be plotted across time for each condition. To assist in developing a larger trial, an effect size will be calculated at post-treatment to describe the standardized difference between conditions. All participants who are randomized and complete a baseline assessment will be included in our analysis. Evaluation of measurement feasibility will focus primarily on descriptive statistics (e.g., frequencies of missing/ incomplete measures). Recruitment and retention over the study duration will be plotted based on the number of participants enrolled into the study and compared to the anticipated rate of recruitment. Veteran feedback on the acceptability of E-PST and treatment satisfaction will be analyzed using rapid qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veteran
* history of mild Traumatic Brain Injury and persistent post-concussion-like symptoms of 3 months
* Brief Symptom Inventory-18 (BSI-18) T-score > 53
* enrolled in VA primary care (appointment within last 12 months)
* English speaking, able to read and write, and able to comprehend study materials

Exclusion Criteria:

* prior, current, or pending enrollment in a cognitive rehabilitation program or other specific TBI intervention program
* moderate to severe TBI or other major neurocognitive disorder
* psychotic disorder, e.g.: schizophrenia spectrum disorder, delusional disorder, schizotypal personality disorder, bipolar or depressive disorder with psychotic features
* acute suicidal ideation
* inpatient psychiatric hospitalization within the past 12 months
* any other illness or condition that would preclude or predictably influence ability to travel to, or engage in, study visits, as determined by the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. King, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Time Frame: Requests will be considered beginning 6 months after final publication.
Access Criteria: Limited datasets in machine-readable electronic format will be created and shared pursuant to a Data Use Agreement (DUA). Appropriate use of the electronic dataset will be specified, as will prohibitions against identifying or re-identifying (i.e., taking steps to identify or re-identify) any individual whose data are included in the dataset.

REFERENCES:
- [Background] King PR Jr, Beehler GP, Donnelly K, Funderburk JS, Wray LO. A Practical Guide to Applying the Delphi Technique in Mental Health Treatment Adaptation: The Example of Enhanced Problem-Solving Training (E-PST). Prof Psychol Res Pr. 2021 Aug;52(4):376-386. doi: 10.1037/pro0000371. Epub 2021 Jun 10. PMID 34446984
- [Background] King PR, Beehler GP, Donnelly K, Funderburk JS, Pengelly C, Wade M, Kretzmer T, Wray LO. Feasibility and acceptability of a brief intervention to improve mild traumatic brain injury recovery: Problem-solving training-concussion. Rehabil Psychol. 2023 May;68(2):135-145. doi: 10.1037/rep0000486. Epub 2023 Mar 9. PMID 36892882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 non-randomized (open trial) participants were enrolled to gather feasibility and acceptability data before randomizing 38 participants to E-PST or HLM control.
Groups:
- E-PST (Randomized): Enhanced Problem-Solving Training (E-PST) randomized arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
  Enhanced Problem-Solving Training (E-PST): E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
- Control (Randomized): Healthy Living Messages (Control) randomized arm. Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
  Healthy Living Messages: Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
- E-PST (Non-randomized): Enhanced Problem-Solving Training (E-PST) non-randomized arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Participants in this open label arm provided feasibility and acceptability data on treatment components. Limited clinical data were collected.
  Enhanced Problem-Solving Training (E-PST): E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
Period: Overall Study
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
Started | 19 | 19 | 12
Completed | 16 | 14 | 7
Not Completed | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- E-PST (Randomized): Enhanced Problem-Solving Training (E-PST) arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Randomized participants were assigned 1:1 to E-PST or HLM.
  Enhanced Problem-Solving Training (E-PST): E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
- Control (Randomized): Healthy Living Messages (Control) arm. Healthy Living Messages (HLM) are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care. Randomized participants were assigned 1:1 to E-PST or HLM.
  Healthy Living Messages: Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
- E-PST (Non-randomized): Enhanced Problem-Solving Training (E-PST) arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training. Non-randomized participants were assigned to E-PST only.
  Enhanced Problem-Solving Training (E-PST): E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
- Total: Total of all reporting groups
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized) | Total
Number analyzed (Participants) | 19 | 19 | 12 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 11 | 48
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.7) | 42 (7.9) | 41 (11.4) | 42 (8.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17 | 17 | 12 | 46
  Female | 2 | 1 | 0 | 3
  Prefer Not to Answer | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 4
  Not Hispanic or Latino | 18 | 16 | 12 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 18 | 18 | 12 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 12 | 50

OUTCOME MEASURES:

1. Primary Outcome: Brief Symptom Inventory-18 (BSI-18) Global Severity Index T-Score
Description: The BSI-18 is a brief measure of psychological distress brought about by common somatic and affective symptoms. It has been validated for use in patients with history of TBI and is appropriate for use in primary care. Similar to a previous trial of PST for mTBI, its Global Severity Index (GSI) T-score will serve as the primary outcome measure. The T-score indicates the number of standard deviations away from the mean. A T-score of 50 is equal to the mean of a reference population (i.e., healthy, sex-matched individuals) with a standard deviation of 10. GSI T-scores range from 30-80, with lower scores signaling an overall lower level of psychological distress.
Time Frame: Up to 24 weeks
Population: All participants
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Control (Randomized): Healthy Living Messages (Control) arm. Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care. Randomized participants were assigned 1:1 to E-PST or HLM.
  Healthy Living Messages: Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
Number analyzed (Participants) | 19 | 19 | 12
units on a scale
  Baseline | 64.21 (2.05) | 65.26 (2.05) | 66.8 (7.9)
  12 Weeks: number analyzed (Participants) | 16 | 15 | 7
  12 Weeks | 61.35 (2.14) | 61.11 (2.17) | 57.0 (8.3)
  24 Weeks: number analyzed (Participants) | 16 | 14 | 0
  24 Weeks | 60.85 (2.14) | 61.83 (2.20) |
Statistical Analysis 1: Comparison: E-PST (Randomized); Test type: Superiority; p = .04, Mixed Models Analysis — 0:24 weeks
Statistical Analysis 2: Comparison: Control (Randomized); Test type: Superiority; p = .05, Mixed Models Analysis — 0:24 weeks
Statistical Analysis 3: Comparison: E-PST (Randomized) vs Control (Randomized); Test type: Superiority; p = .58, Mixed Models Analysis — 12:12 weeks

2. Secondary Outcome: Applied Cognition-General Concerns-Short Form (ACGC-8a)
Description: An 8-item checklist of general cognitive concerns over the past week. Items were generated and validated as part of the National Institute of Health's Patient-Reported Outcome Measurement Information System (PROMIS). Raw scores are converted to T-scores (range = 23.3-62.7), with higher scores signaling relatively fewer cognitive concerns. The T-score indicates the number of standard deviations away from the mean. A T-score of 50 is equal to the mean of a reference population (i.e., healthy individuals) with a standard deviation of 10.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- E-PST: Enhanced Problem-Solving Training (E-PST) arm. E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
  Enhanced Problem-Solving Training (E-PST): E-PST is a combined treatment that is comprised of brief problem-solving training and compensatory cognitive skills training.
- Control: Healthy Living Messages (Control) arm. Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
  Healthy Living Messages: Healthy Living Messages are primary care-congruent messages that consist of simple advice regarding general health behaviors and preventive care.
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 40.44 (1.71) | 44.47 (1.71)
  12 Weeks: number analyzed (Participants) | 16 | 15
  12 Weeks | 38.94 (1.80) | 40.80 (1.83)
  24 Weeks: number analyzed (Participants) | 16 | 14
  24 Weeks | 40.66 (1.80) | 44.95 (1.86)

3. Secondary Outcome: Applied Cognition-Abilities-Short Form (ACA-8a)
Description: An 8-item checklist of self-perceived cognitive abilities over the past week, developed as part of the National Institute of Health's Patient-Reported Outcome Measurement Information System (PROMIS). Raw scores are converted to T-scores (range = 27-64.8) with higher scores signaling higher perceived cognitive abilities. The T-score indicates the number of standard deviations away from the mean. A T-score of 50 is equal to the mean of a reference population (i.e., healthy individuals) with a standard deviation of 10.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 43.16 (1.65) | 41.52 (1.65)
  12 Weeks: number analyzed (Participants) | 16 | 15
  12 Weeks | 44.06 (1.75) | 42.50 (1.78)
  24 Weeks: number analyzed (Participants) | 16 | 14
  24 Weeks | 44.46 (1.74) | 39.00 (1.82)

4. Secondary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: A brief test of verbal learning, recall, and recognition. Participants are read a word list over 3 learning trials, and are asked to recall as many words as possible after a 25-minute delay. Raw scores are converted to T-scores (range = 20 to 80), with higher scores signaling better verbal memory performance. The T-score indicates the number of standard deviations away from the mean. A T-score of 50 is equal to the mean of a reference population (i.e., healthy, age-matched individuals) with a standard deviation of 10.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline- Delayed Recall T-Score | 34.11 (2.66) | 38.12 (2.70)
  12 Weeks- Delayed Recall T-Score: number analyzed (Participants) | 16 | 15
  12 Weeks- Delayed Recall T-Score | 38.19 (2.82) | 35.99 (2.88)
  24 Weeks- Delayed Recall T-Score: number analyzed (Participants) | 16 | 14
  24 Weeks- Delayed Recall T-Score | 33.88 (2.82) | 35.44 (2.94)

5. Secondary Outcome: Wechsler Adult Intelligence Scale- Fourth Edition (WAIS-IV) Digit Span
Description: A brief verbal attention test. Participants are presented with a sequence of digits and asked to repeat them forward and backward. Raw scores are converted to scaled scores (range = 1-19) with corresponding percentile ranks (range = 1 to 99); higher scaled scores and percentile ranks signal better overall performance.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 19
score on a scale
  Baseline | 7.16 (0.35) | 6.95 (0.35)
  12 Weeks: number analyzed (Participants) | 16 | 15
  12 Weeks | 7.47 (0.37) | 7.10 (0.37)
  24 Weeks: number analyzed (Participants) | 16 | 14
  24 Weeks | 7.72 (0.37) | 7.06 (0.38)

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: A 9-item measure of cognitive, affective, and somatic depressive symptoms validated for use in primary care. Scores range from 0 to 27, with lower scores signaling lower mood symptoms.
Time Frame: Up to 24 weeks
Population: All participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
Number analyzed (Participants) | 19 | 19 | 12
units on a scale
  Baseline | 11.95 (1.32) | 11.95 (1.32) | 11.7 (6.7)
  12 Weeks: number analyzed (Participants) | 16 | 15 | 7
  12 Weeks | 10.57 (1.38) | 11.07 (1.39) | 8.6 (6.7)
  24 Weeks: number analyzed (Participants) | 16 | 14 | 0
  24 Weeks | 8.82 (1.38) | 12.24 (1.41) |

7. Secondary Outcome: PTSD Checklist for DSM-5 (PCL5)
Description: A 20-item measure of DSM-5 symptoms related to trauma, organized over re-experiencing, avoidance, hyperarousal, and cognitive/mood domains. Score range from 0-80, with lower scores signaling less severe PTSD symptoms.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
Number analyzed (Participants) | 18 | 15 | 12
units on a scale
  Baseline | 31.15 (4.80) | 27.90 (5.19) | 40.3 (17.9)
  12 Weeks: number analyzed (Participants) | 16 | 13 | 7
  12 Weeks | 31.04 (5.00) | 28.67 (5.43) | 35.3 (18.9)
  24 Weeks: number analyzed (Participants) | 14 | 13 | 0
  24 Weeks | 24.52 (5.20) | 30.30 (5.43) |

8. Secondary Outcome: Alcohol Use Disorders Identification Test-Consumption Questions (AUDIT-C)
Description: A 3-item measure of the frequency and severity of alcohol intake over the past year. Scores range from 0 to 12, with lower scores signaling less overall alcohol consumption.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 17 | 19
units on a scale
  Baseline | 2.90 (0.62) | 4.37 (0.61)
  12 Weeks: number analyzed (Participants) | 15 | 15
  12 Weeks | 2.37 (0.63) | 4.21 (0.63)
  24 Weeks: number analyzed (Participants) | 16 | 14
  24 Weeks | 1.95 (0.63) | 4.00 (0.64)

9. Secondary Outcome: Brief Addictions Monitor-Revised (BAM-R)
Description: A 17-item measure of substance misuse and associated functional impairment. The Use subscale score ranges from 0-12, with lower scores signaling no (0) or relatively lower substance use.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 12 | 15
units on a scale
  Baseline | 2.47 (0.65) | 3.02 (0.59)
  12 Weeks: number analyzed (Participants) | 9 | 13
  12 Weeks | 2.69 (0.72) | 3.91 (0.61)
  24 Weeks: number analyzed (Participants) | 8 | 11
  24 Weeks | 2.39 (0.75) | 3.73 (0.65)

10. Secondary Outcome: Pain Symptom Survey (PEG)
Description: A 3-item pain assessment that has been validated for use in VA patients. Respondents are asked to report their average level of pain, the average impact of pain on their ability to enjoy life, and the average level of interference on daily activities on a scale of 0 to 10. Ratings on each domain are averaged to calculate a composite score, which ranges from 0 to 10, with lower scores signaling lower overall pain.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 5.28 (0.51) | 5.56 (0.51)
  12 Weeks: number analyzed (Participants) | 16 | 15
  12 Weeks | 5.36 (0.54) | 4.89 (0.55)
  24 Weeks: number analyzed (Participants) | 16 | 14
  24 Weeks | 4.67 (0.54) | 4.74 (0.56)

11. Secondary Outcome: Patient Global Impressions of Change (PGIC)
Description: A 7-point single-item rating scale that asks patients to rate their overall impression of response to treatment. Ratings range from "no change" to "a great deal better." Ratings range from 0 to 7, with higher ratings signaling greater perceived change in response to treatment. Because ratings are only collected after receiving a given treatment, baseline values are not collected.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 16 | 15
units on a scale
  12 weeks | 4.19 (0.44) | 2.87 (0.46)
  24 weeks: number analyzed (Participants) | 16 | 14
  24 weeks | 4.19 (0.47) | 2.92 (0.51)

12. Secondary Outcome: World Health Organization Quality of Life - BREF (WHOQOL-BREF)
Description: A 26-item abbreviated version of the full-length WHOQOL measure that evaluates disability and quality of life in domains such as social relationships, physical and mental health, and satisfaction with person-environment interactions. Raw scores are averaged to compute domain scores (range = 4-20), with higher scores signaling an overall higher quality of life.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST | Control
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline- Physical | 12.66 (0.59) | 13.23 (0.59)
  12 weeks- Physical: number analyzed (Participants) | 16 | 15
  12 weeks- Physical | 12.21 (0.62) | 13.40 (0.64)
  24 weeks- Physical: number analyzed (Participants) | 16 | 14
  24 weeks- Physical | 12.86 (0.62) | 12.57 (0.65)
  Baseline- Psychological | 13.02 (0.71) | 13.05 (0.71)
  12 weeks- Psychological: number analyzed (Participants) | 16 | 15
  12 weeks- Psychological | 13.35 (0.74) | 12.59 (0.75)
  24 weeks- Psychological: number analyzed (Participants) | 16 | 14
  24 weeks- Psychological | 13.18 (0.74) | 11.83 (0.76)
  Baseline- Social | 12.63 (0.84) | 15.02 (0.84)
  12 weeks- Social: number analyzed (Participants) | 16 | 15
  12 weeks- Social | 12.43 (0.87) | 14.64 (0.88)
  24 weeks- Social: number analyzed (Participants) | 16 | 14
  24 weeks- Social | 13.18 (0.87) | 13.98 (0.90)
  Baseline- Environment | 15.82 (0.46) | 16.39 (0.46)
  12 weeks- Environment: number analyzed (Participants) | 16 | 15
  12 weeks- Environment | 15.41 (0.49) | 16.50 (0.50)
  24 weeks- Environment: number analyzed (Participants) | 16 | 14
  24 weeks- Environment | 15.83 (0.49) | 16.12 (0.51)

13. Other Pre Specified Outcome: Neurobehavioral Symptom Inventory
Description: A 22-item checklist of affective, cognitive, and somatosensory symptoms commonly reported after concussion. Scores range from0 to 88, with lower scores signaling lower overall symptom reports.
Time Frame: Up to 24 weeks
Population: Randomized participants
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
Number analyzed (Participants) | 19 | 19 | 12
units on a scale
  Baseline | 42.42 (3.59) | 41.42 (3.59) | 43.3 (17.2)
  12 weeks: number analyzed (Participants) | 16 | 15 | 7
  12 weeks | 40.35 (3.70) | 38.02 (3.74) | 35.3 (17.4)
  24 weeks: number analyzed (Participants) | 16 | 14 | 0
  24 weeks | 37.79 (3.70) | 38.81 (3.78) |

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | E-PST (Randomized) | Control (Randomized) | E-PST (Non-randomized)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/19 | 0/12
Other Adverse Events (participants affected / at risk) | 8/19 | 6/19 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-PST (Randomized) (N=19) | Control (Randomized) (N=19) | E-PST (Non-randomized) (N=12)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | NA — Strain/sprain or contusion
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-PST (Randomized) (N=19) | Control (Randomized) (N=19) | E-PST (Non-randomized) (N=12)
Emotional distress, depression (Psychiatric disorders) | 6 (6) | 6 (7) | 0 (0)
COVID (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Positive COVID-19 diagnosis, respiratory symptoms
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study emphasized feasibility and acceptability metrics. Given the small number of participants enrolled in the randomized pilot trial, there was not sufficient power to robustly detect clinical effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT03759223/Prot_SAP_ICF_000.pdf